CLINICAL TRIAL: NCT00727636
Title: Pilot Study of Immunogenicity and Tolerability to the Quadrivalent Human Papillomavirus Virus-like Particle (VLP) Vaccine (Gardasil) Among IBD Patients on Immunosuppressive Therapy Compared to Healthy Children and Youth Adult Females
Brief Title: Immunogenicity to Human Papillomavirus Vaccine (Gardasil) Among IBD Patients on Immunosuppressive Therapy
Acronym: HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Athos Bousvaros, MD, Children's Hospital Boston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 07-09-0344
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Results first posted 2011-05-27 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Inflammatory Bowel Disease
Keywords: inflammatory bowel disease (IBD); immunogenicity; safety; HPV; Gardasil; vaccine
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gardasil vaccine - Prospective Study (Experimental): Prospective study participants received the Gardasil vaccine during the study
  Interventions: Biological: Gardasil vaccine
- Retrospective Study (No Intervention): Retrospective study participants had blood drawn in the study after they had received the Gardasil vaccine from their primary medical provider

INTERVENTIONS:
Biological: Gardasil vaccine — standard 0.5 mL dose of Gardasil vaccine given at Day 0, Month 2, and Month 6
  Other Names: Gardasil, HPV vaccine
  Arms: Gardasil vaccine - Prospective Study

SUMMARY:
Many IBD patients take immunosuppressive agents and we are uncertain as to their capacity to mount a truly protective response after vaccination. If IBD patients do not have an adequate immunological response, they may need to increase the dosage or get booster shots. Many clinicians who treat patients with autoimmune diseases are asking if the vaccine is safe and effective. Thus, this study has important clinical and public health significance because more than one million people in the United States have been diagnosed with IBD.

There is not much studied about HPV and immunocompromised patients. Research on healthy women who were immunized with a set of three HPV vaccines demonstrated significantly increased antibody titers. In addition, they had significantly reduced HPV incident and persistent infection and HPV-related disease (cervical, vulvar, and vaginal cancers, cervical intraepithelial neoplasia, genital warts) through five years of follow-up compared to controls who received a placebo. The HPV vaccine was well tolerated without significant side effects.

The aims of this research are to measure the immune response in 9-26 year old IBD patients who are on immunosuppressive agents after receiving the HPV vaccine compared with historical controls. We will also evaluate the number and type of vaccine-associated adverse events as well as the disease activity and flare-ups that occur after each dose of vaccine. We hypothesize that IBD patients on immunosuppressive therapy will have have a similar immune response to HPV types 6, 11, 16 and 18 at one month postdose 3 compared to healthy age-matched historical controls.

The patient population includes IBD patients who are on immunosuppressive medications. Recruiting approximately 100 patients will provide adequate power for the study. A blood sample will be taken from all IBD patients to evaluate baseline antibody levels and markers (e.g., ESR, CBC, albumin) before or immediately after immunization with the HPV vaccine. Lab tests will be redrawn at 7 months to evaluate the level of antibody titers and follow the markers. During the study, we will track basic laboratory measures, disease status by using the Pediatric Crohn's Disease Active Index or Harvey-Bradshaw Index for UC, side effects from the vaccinations, and other adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Crohn's disease, ulcerative colitis, or indeterminate colitis diagnosed by standard clinical, radiographic, endoscopic, and histologic criteria.
2. Actively followed by a physician at the Children's' Hospital gastroenterology (GI) or IBD Center, or patient is referred by local clinic or hospital for our study.
3. Female gender
4. Age 9-26 years
5. Patient (18 years old) or parent is willing to provide informed consent.
6. Is currently on an immunomodulator and/or TNF inhibitor for ≥ 30 days prior to enrollment. Patients may also be using prednisone or aminosalicylates in addition to the immunomodulator or TNF inhibitor. Standard concomitant medications (e.g. antibiotics, antihistamines, acetaminophen) will be allowed

Exclusion Criteria:

1. Male gender
2. Unwilling to provide consent
3. New immunomodulator added within the last 30 days, and was not previously on any immunomodulator
4. History of bleeding disorder that would make hematoma likely (e.g., hemophilia, von Willebrand's disease) or on anti-coagulation therapy (certain cases may be allowed; each case will be assessed by study doctor)
5. Hypersensitivity to the ingredients/components of the vaccine (e.g., aluminum, yeast)
6. Known pregnancy or positive pregnancy test. We will obtain a urinary pregnancy test before each dose of the vaccine is administered. Subjects participating will be informed during the consent/assent procedures that the safety of this vaccine has not been proven in pregnant women, and will be advised not to become pregnant during the study and counseled according to the guidelines of the Children's Hospital IRB.
7. Previously received HPV vaccination.

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athos Bousvaros, MD, Principal Investigator — Boston Children's Hospital; Denise L Jacobson, PhD, MPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location - Children's Hospital Boston, including Waltham Infusion Center, and Maine Medical Center. Patients were recruited during a scheduled clinical or Remicade infusion visit, a hospital admission, by contact through mail followed by a phone call, or through referral from local hospitals. Recruitment period -April 2008 through April 2010
Groups:
- Prospective Cohort: Received Gardasil as part of study
- Retrospective Cohort: Patients received Gardasil vaccine from their primary medical provider. They had blood drawn for the study after they completed the vaccine
Period: Overall Study
Arm/Group | Prospective Cohort | Retrospective Cohort
Started | 37 | 15
Completed | 33 | 15
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective Cohort | Retrospective Cohort | Total
Number analyzed (Participants) | 37 | 15 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 6 | 39
  Between 18 and 65 years | 4 | 9 | 13
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 14.9 (3.1) | 18.9 (3.5) | 16.1 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 15 | 52
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 15 | 52

OUTCOME MEASURES:

1. Primary Outcome: Antibody Titer to HPV 6
Time Frame: Month 7
Measure: Geometric Mean (95% Confidence Interval); unit: milli-Merck units/mL
Arm/Group | Prospective Cohort | Retrospective Cohort
Number analyzed (Participants) | 33 | 15
milli-Merck units/mL | 1079.9 [783 to 1489.3] | 173.4 [91.3 to 329.5]

2. Primary Outcome: Antibody Titer to HPV 11
Time Frame: Month 7
Population: Number of participants who completed all vaccine doses
Measure: Geometric Mean (95% Confidence Interval); unit: milli-Merck units/mL
Arm/Group | Prospective Cohort | Retrospective Cohort
Number analyzed (Participants) | 33 | 15
milli-Merck units/mL | 1681.8 [1189.9 to 2377.2] | 267.3 [122.4 to 583.8]

3. Primary Outcome: Antibody Titers to HPV 16
Description: Geometric mean titer (95% CI)
Time Frame: Month 7
Measure: Geometric Mean (95% Confidence Interval); unit: milli-Merck units/mL
Arm/Group | Prospective Cohort | Retrospective Cohort
Number analyzed (Participants) | 33 | 15
milli-Merck units/mL | 3975.1 [2492.2 to 6340.6] | 802.7 [391.1 to 1676.6]

4. Primary Outcome: Antibody Titer to HPV 18
Description: Geometric mean titer (95%CI)
Time Frame: Month 7
Measure: Geometric Mean (95% Confidence Interval); unit: milli-Merck units/mL
Arm/Group | Prospective Cohort | Retrospective Cohort
Number analyzed (Participants) | 33 | 15
milli-Merck units/mL | 857.6 [472.4 to 1556.6] | 79.5 [26.3 to 240.5]

ADVERSE EVENTS:
Time Frame: From the 1st dose of vaccine until 1 month after the 3rd dose of vaccine
Description: Adverse events were only evaluated in the Prospective Study patients. The Retrospective Study patients were not given the vaccine as part of this study.
Arm/Group | Prospective Cohort | Retrospective Cohort
Serious Adverse Events (participants affected / at risk) | 5/37 | 0/0
Other Adverse Events (participants affected / at risk) | 11/37 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospective Cohort (N=37) | Retrospective Cohort (N=0)
Admitted to hospital (Gastrointestinal disorders) | 2 (2) | 0 (0) — exacerbation of inflammatory bowel disease
Admitted to hospital (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — pneumonia
Admitted to hospital (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Endometriosis with an ovarian torsion
Went to emergency department (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Sinus pain
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospective Cohort (N=37) | Retrospective Cohort (N=0)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asthma related symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rectal bleeding and diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Axillary abscess (General disorders) | 1 (1) | 0 (0)
Rash on their chin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal pain (General disorders) | 3 (3) | 0 (0)
Migraine (General disorders) | 1 (1) | 0 (0)
Swelling and severe pain in arm (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less